CLINICAL TRIAL: NCT06611345
Title: A Single-Arm, Phase 1b Study to Assess Tumor-Treating Fields (TTF) in Combination With Durvalumab and Gemcitabine/Cisplatin (GemCis) as the First-Line Treatment of Unresectable Biliary Tract Cancers (BTC)
Brief Title: A Study of Tumor-Treating Fields in Combination With Durvalumab and Gemcitabine/Cisplatin in Biliary Tract Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Healthy Life Innovation Medical Technology Co., Ltd (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-07
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Biliary Tract Cancers (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tumor Treating Fields combined with durvalumab and GemCis (Experimental)
  Interventions: Device: Tumor Treating Fields; Drug: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Device: Tumor Treating Fields — Tumor treating fields will be used each day.
Drug: Durvalumab — Durvalumab 1500 mg will be administrated via Intravenous (IV) infusion Once Every 3 weeks (Q3W) on day 1 of each cycle for up to 8 cycles. And then 1500 mg Once Every 4 weeks (Q4W) on day 1 of each cycle until confirmed progressive disease (PD).
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 will be given on Days 1 and 8 of each cycle up to 8 cycles.
Drug: Cisplatin — Cisplatin 25 mg/m2 will be given on Days 1 and 8 of each cycle up to 8 cycles.

SUMMARY:
Unresectable BTC represents an area of unmet medical need due to its very aggressive nature, limited treatment options, and poor prognosis. This study is to evaluate the efficacy and safety of adding TTF to the established regimen of durvalumab plus GemCis for the treatment of patients with previously untreated, unresectable BTC.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial.
2. Male or female patients between the ages of 18 and 75 years (including 18 and 75 years).
3. Body weight > 30 kg.
4. Histologically confirmed, unresectable adenocarcinoma of the biliary tract, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma.
5. Patients with the previously untreated disease if unresectable or metastatic at initial diagnosis will be eligible.
6. Patients with recurrent disease >6 months after curative surgery or >6 months after the completion of adjuvant therapy (chemotherapy and/or radiation) will be eligible (but he/she does not receive systemic treatment as the first-line therapy).
7. At least 1 measurable lesion that qualifies as a RECIST 1.1 Target Lesion (TL) at baseline.
8. ECOG PS of 0 or 1.
9. Life expectancy ≥12 weeks at the time of screening.
10. No prior exposure to immune-mediated therapy, including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines.
11. Patients must have adequate organ function as indicated by the following laboratory values: Hemoglobin ≥9.0 g/dL; Absolute neutrophil count ≥1.5 ×109/L; Platelet count ≥100 ×109/L. No blood transfusion, granulocyte colony-stimulating factor (G-CSF), filgrastim and other drugs are used within 2 weeks before the examination. Serum bilirubin ≤2.0 × the upper limit of normal (ULN); This will not apply to patients with confirmed Gilbert's syndrome. Any clinically significant biliary obstruction should be resolved before treatment. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤5 × ULN. Creatinine clearance (CL) >50 mL/min per 24-hour urine or as calculated by Cockroft and Gault formula (using actual body weight).
12. Patients (women of childbearing potential and males with fertile female partners) must be willing to use the currently accepted reliable contraception method from the time of screening throughout the total duration of the study treatment and the drug washout period (180 days after the last dose of GemCis or 90 days after the last dose of durvalumab monotherapy). These measures include, but are not limited to, oral or implantable injections of hormonal contraceptives; intrauterine birth control ring or placement of IUS intrauterine device); or use of barrier methods such as condoms or septum and spermicide products. Postmenopausal women over 50 years of age must have been amenorrheic for at least 12 months to be considered non-childbearing potential.
13. Patients with HBV infection (as characterized by positive hepatitis B surface antigen [HBsAg] and/or anti-hepatitis B core antibodies (anti-HBc) with detectable HBV deoxyribonucleic acid (DNA) [above the limit of detection per local laboratory]) must receive antiviral therapy prior to treatment per institutional practice to ensure adequate viral suppression. Patients must remain on antiviral therapy for the study duration and for 6 months after the last dose of study treatment. Patients who test positive for anti-HBc with undetectable HBV DNA (under the limit of detection per local laboratory) do not require antiviral therapy unless HBV DNA reaches detectable limits per local laboratory during the course of treatment. Patients with active co-infection of HBV and HCV as evidenced by positive anti-HCV antibody and actively co-infected with HBV and hepatitis D virus are not eligible.
14. Able to operate TTF device independently or with the help of a caregiver.

Exclusion Criteria:

1. Patients previously received systemic treatment as the first-line therapy.
2. Ampullary carcinoma.
3. History of allogeneic organ transplantation.
4. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: Patients with vitiligo or alopecia; Patients with hypothyroidism (e.g., following Hashimoto syndrome) are stable on hormone replacement; Any chronic skin condition that does not require systemic therapy; Patients without active disease in the last 5 years may be included but only after consultation with the investigator/ Study Physician; Patients with celiac disease controlled by diet alone.
5. Uncontrolled intercurrent illness, including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase the risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
6. History of another primary malignancy, except for: Malignancy was treated with curative intent and with no known active disease ≥5 years before the first dose of the investigational product (IP) and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; Adequately treated carcinoma in situ without evidence of disease.
7. History of leptomeningeal carcinomatosis.
8. History of active primary immunodeficiency.
9. Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), or human immunodeficiency virus (positive HIV 1/2 antibodies).
10. Any unresolved toxicity NCI CTCAE Grade ≥2 from a previous anticancer therapy, with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
11. Brain metastases or spinal cord compression (including asymptomatic and adequately treated disease). Patients with suspected brain metastases at screening should have an MRI (preferred) or CT scan, each preferably with IV contrast of the brain prior to study entry.
12. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
13. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
14. Radiation therapy, including palliative radiation, is not allowed before the study, with an exception of radiation given in an adjuvant setting.
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note that patients, if enrolled, should not receive a live vaccine while receiving IP and up to 30 days after the last dose of IP.
16. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note that minor surgery of isolated lesions for palliative intent is acceptable if performed more than 14 days prior to the first dose of IP.
17. Patients who have received prior immune-mediated therapy, including, but not limited to, other anti-PD-1, anti-PD-L1, or anti-CTLA-4.
18. Prior locoregional therapy such as radioembolization.
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion: Intranasal, inhaled, or topical steroids, or local steroid injections (e.g., intra-articular injection); Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
20. Participation in another clinical study with an IP administered in the last 3 months.
21. Previous IP assignment in the present study.
22. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
23. Prior randomization or treatment in a previous durvalumab clinical study, regardless of treatment arm assignment.
24. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to use effective birth control from screening to 180 days after the last dose of GemCis or 90 days after the last dose of durvalumab monotherapy.
25. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
26. Active infection of hepatitis C as evidenced by detectable HCV RNA per local laboratory. Patients who test positive for hepatitis C (HCV) antibody may be enrolled if HCV RNA is undetectable.
27. Known allergy or hypersensitivity to medical adhesives or hydrogel.
28. Implantable electronic medical devices such as cardiac pacemakers.
29. Metallic medical devices, such as bone nails, were implanted in the chest and abdomen.
30. Patients with infection, ulcer or unhealed wound at the electrode application site.
31. Patients with symptomatic ascites, pleural effusion, pericardial effusion, etc., unless the condition is well controlled after clinical treatment (including therapeutic puncture).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months after the enrollment of the last patient.
  PFS is defined as the time from the date of treatment until the date of Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)-defined radiological PD or death.

SECONDARY OUTCOMES:
Safety profile | Up to 24 months after the enrollment of the last patient.
  Safety profile is defined as the incidence, frequency and severity of adverse events (AEs) noted in patients treated with study treatments.
Objective response rate (ORR) | Up to 24 months after the enrollment of the last patient.
  ORR is defined as the number (%) of patients with at least 1 visit response of complete response (CR) or partial response (PR).
Disease control rate (DCR) | Up to 24 months after the enrollment of the last patient.
  DCR is defined as the rate of best objective response of CR, PR, or stable disease (SD).
Duration of response (DOR) | Up to 24 months after the enrollment of the last patient.
  DOR is defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression.
Overall survival (OS) | Up to 24 months after the enrollment of the last patient.
  OS is defined as the time from the date of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, China

IPD SHARING:
Plan to Share IPD: No